CLINICAL TRIAL: NCT03148834
Title: A Randomized Study to Evaluate Controlled Reperfusion With Venous Blood and Dextran for Myocardial Protection Compared With Standard Angioplasty During Primary Angioplasty in Patients With Acute Myocardial Infarction and TIMI 0/1 Flow.
Brief Title: Dextran Use for Primary Angioplasty Protection in Acute Myocardial Infarction
Acronym: DUPAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Cardiovascular Salta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 052017
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Acute Myocardial Infarction With ST Elevation
Keywords: Acute Myocardial Infarction Reperfusion Injury
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Reperfusion Primary Angioplasty (Experimental): Patients admitted with acute myocardial infarction and TIMI flow 0/1, will be treated with the use of an intracoronary venous blood solution and dextran to protect the myocardium during reperfusion.
  Interventions: Procedure: Controlled Reperfusion
- Standard Primary Coronary Angioplasty (No Intervention): Patients admitted with an acute myocardial infarction and TIMI flow 0/1, will be treated with primary angioplasty according to norms described in the international guidelines of treatment.

INTERVENTIONS:
Procedure: Controlled Reperfusion — Patients will be treated in the occluded coronary with a solution of venous blood and Dextran, prior to the Stenting procedure.
  Controlled Reperfusion PCI consists of crossing the culprit lesion with guidewire and then advancing a balloon (over the wire) to the distal segment of the culprit vessel. Proximal to the main distal branch, inflate the balloon to low atmospheres, remove the guide wire and inject the solution through the light of the balloon. Then reposition the guidewire, perform angioplasty as usual on the lesion. If there is a large residual thrombus load and at the operator's discretion, change the balloon by a manual thromboaspiration catheter and use it.
  Then perform stenting of the lesion. The solution will be given with a 1 cc syringe as a slow bolus, controlling symptoms and ST segment response.
  The compounds in solution are venous blood drawn from the patient after administration of heparin and mixed with dextran in a 3/1 ratio.
  Arms: Control Reperfusion Primary Angioplasty

SUMMARY:
Reperfusion therapy in acute myocardial infarction saves viable myocardium, but paradoxically reestablishment of coronary artery flow also induces damage and cell death, decreasing the full benefit of reperfusion in terms of reduction of infarct size and preservation of ventricular function . Myocardial reperfusion can in itself produce more damage and cell death, this process defines the phenomenon of reperfusion injury, which could be prevented by applying additional therapies.

DETAILED DESCRIPTION:
During myocardial ischemia, due to lack of O2, the myocyte leaves energy production from the aerobic metabolism of lipids and the production of energy in the form of phosphates will depend, in this situation, on the anaerobic metabolism of glucose. As a result they are consumed muscle glycogen stores that produce little ATP, and also generating acidosis. The cell membrane loses its ability to maintain the fluid's electrolyte balance. Cellular edema is generated by the entry of sodium and water, leading to cell rupture. During ischemia and reperfusion free radicals are produced that stimulate inflammation and consequently release prothrombotic and cytotoxic substances that also produce cellular damage. Due to its osmotic, antithrombotic, anti-inflammatory and rheological effects, dextran could be useful in this scenario.

The administration of a solution in the distal bed, for the protection of the myocardium, before opening the epicardial artery is called by us "controlled reperfusion". The researchers think, using a solution with venous blood, containing less O2 but retaining buffer properties; enriched with Dextran, which has onctic power, anti-inflammatory and anticoagulant properties, and molecules similar to glucose; results in a potentially useful solution for myocardial protection in this scenario.

The group of investigators expect that controlled reperfusion treatment will reduce the incidence of ST correction and infarct size by 20-30%, improving the prognosis in terms of mortality and heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Women and men over 18 years of age
* First acute myocardial infarction with ST elevation, within 6 hours of the initial symptoms, that are admitted for primary PCI at the Hospital San Bernardo.
* TIMI 0 or 1 flow in the culprit artery.

Exclusion Criteria:

* Not able or willing to give informed consent.
* Participate in another protocol.
* Pregnancy.
* History of any of the diseases listed: cardiomyopathy, valvular disease severe, any disease with a life expectancy of less than 1 year.
* Contraindication for protocol drugs (Dextran).
* LBBB or pacemaker.
* Prolonged cardiopulmonary resuscitation.
* Cardiogenic shock.
* Left main coronary lesion or culprit lesion in venous graft.
* Large artery not feasible for PCI, guilty vessel of small caliber or very distal lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in ST segment elevation from baseline | At six hours
  Resolution of ST segment elevation in the EKG
Total Mortality | One year
  Incidence of death

SECONDARY OUTCOMES:
Infarct size | Six month
  With the use of Myocardial Spect Imaging

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steg PG, Dabbous OH, Feldman LJ, Cohen-Solal A, Aumont MC, Lopez-Sendon J, Budaj A, Goldberg RJ, Klein W, Anderson FA Jr; Global Registry of Acute Coronary Events Investigators. Determinants and prognostic impact of heart failure complicating acute coronary syndromes: observations from the Global Registry of Acute Coronary Events (GRACE). Circulation. 2004 Feb 3;109(4):494-9. doi: 10.1161/01.CIR.0000109691.16944.DA. Epub 2004 Jan 26. PMID 14744970
- [Background] Velazquez EJ, Francis GS, Armstrong PW, Aylward PE, Diaz R, O'Connor CM, White HD, Henis M, Rittenhouse LM, Kilaru R, van Gilst W, Ertl G, Maggioni AP, Spac J, Weaver WD, Rouleau JL, McMurray JJ, Pfeffer MA, Califf RM; VALIANT registry. An international perspective on heart failure and left ventricular systolic dysfunction complicating myocardial infarction: the VALIANT registry. Eur Heart J. 2004 Nov;25(21):1911-9. doi: 10.1016/j.ehj.2004.08.006. PMID 15522470
- [Background] Hellermann JP, Jacobsen SJ, Redfield MM, Reeder GS, Weston SA, Roger VL. Heart failure after myocardial infarction: clinical presentation and survival. Eur J Heart Fail. 2005 Jan;7(1):119-25. doi: 10.1016/j.ejheart.2004.04.011. PMID 15642543
- [Background] Campo G, Valgimigli M, Gemmati D, Percoco G, Tognazzo S, Cicchitelli G, Catozzi L, Malagutti P, Anselmi M, Vassanelli C, Scapoli G, Ferrari R. Value of platelet reactivity in predicting response to treatment and clinical outcome in patients undergoing primary coronary intervention: insights into the STRATEGY Study. J Am Coll Cardiol. 2006 Dec 5;48(11):2178-85. doi: 10.1016/j.jacc.2005.12.085. Epub 2006 Nov 13. PMID 17161242
- [Background] Komamura K, Kitakaze M, Nishida K, Naka M, Tamai J, Uematsu M, Koretsune Y, Nanto S, Hori M, Inoue M, et al. Progressive decreases in coronary vein flow during reperfusion in acute myocardial infarction: clinical documentation of the no reflow phenomenon after successful thrombolysis. J Am Coll Cardiol. 1994 Aug;24(2):370-7. doi: 10.1016/0735-1097(94)90290-9. PMID 8034870
- [Background] Karila-Cohen D, Czitrom D, Brochet E, Faraggi M, Seknadji P, Himbert D, Juliard JM, Assayag P, Steg PG. Decreased no-reflow in patients with anterior myocardial infarction and pre-infarction angina. Eur Heart J. 1999 Dec;20(23):1724-30. doi: 10.1053/euhj.1999.1714. PMID 10562480
- [Background] Niccoli G, Lanza GA, Shaw S, Romagnoli E, Gioia D, Burzotta F, Trani C, Mazzari MA, Mongiardo R, De Vita M, Rebuzzi AG, Luscher TF, Crea F. Endothelin-1 and acute myocardial infarction: a no-reflow mediator after successful percutaneous myocardial revascularization. Eur Heart J. 2006 Aug;27(15):1793-8. doi: 10.1093/eurheartj/ehl119. Epub 2006 Jul 7. PMID 16829540
- [Background] Niccoli G, Giubilato S, Russo E, Spaziani C, Leo A, Porto I, Leone AM, Burzotta F, Riondino S, Pulcinelli F, Biasucci LM, Crea F. Plasma levels of thromboxane A2 on admission are associated with no-reflow after primary percutaneous coronary intervention. Eur Heart J. 2008 Aug;29(15):1843-50. doi: 10.1093/eurheartj/ehn325. Epub 2008 Jul 10. PMID 18617477
- [Background] Uyarel H, Cam N, Okmen E, Kasikcioglu H, Tartan Z, Akgul O, Simsek D, Cetin M, Bozbeyoglu E, Buturak A, Uzunlar B. Level of Selvester QRS score is predictive of ST-segment resolution and 30-day outcomes in patients with acute myocardial infarction undergoing primary coronary intervention. Am Heart J. 2006 Jun;151(6):1239.e1-7. doi: 10.1016/j.ahj.2006.03.019. PMID 16781226
- [Background] Buller CE, Fu Y, Mahaffey KW, Todaro TG, Adams P, Westerhout CM, White HD, van 't Hof AW, Van de Werf FJ, Wagner GS, Granger CB, Armstrong PW. ST-segment recovery and outcome after primary percutaneous coronary intervention for ST-elevation myocardial infarction: insights from the Assessment of Pexelizumab in Acute Myocardial Infarction (APEX-AMI) trial. Circulation. 2008 Sep 23;118(13):1335-46. doi: 10.1161/CIRCULATIONAHA.108.767772. Epub 2008 Sep 8. PMID 18779444
- [Background] Bulluck H, Yellon DM, Hausenloy DJ. Reducing myocardial infarct size: challenges and future opportunities. Heart. 2016 Mar;102(5):341-8. doi: 10.1136/heartjnl-2015-307855. Epub 2015 Dec 16. PMID 26674987
- [Background] Hausenloy DJ, Yellon DM. Myocardial ischemia-reperfusion injury: a neglected therapeutic target. J Clin Invest. 2013 Jan;123(1):92-100. doi: 10.1172/JCI62874. Epub 2013 Jan 2. PMID 23281415